CLINICAL TRIAL: NCT03456869
Title: The Application and Clinical Accuracy of Patient-specific Implants in Genioplasty
Brief Title: Clinical Accuracy of Patient-specific Implants in Genioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Xudong Wang, Acting chair of Department of Oral and Craniomaxillofacial Surgery, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSIcmfs03
Record Dates: First submitted 2018-02-05; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Genioplasty; Chin Microgenia; Chin Macrogenia
Keywords: patient specific implant; computer-aided surgery; clinical accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSI group (Experimental): The patient specific implant (PSI) is used to completed the genioplasty.
  Interventions: Device: Patient Specific Implant

INTERVENTIONS:
Device: Patient Specific Implant — The patient specific implant is used to simultaneously complete the reposition and fixation of the chin.

SUMMARY:
The purpose of this study is to assess the accuracy and clinical validation of patient specific implants (PSI) technique for genioplasty.

DETAILED DESCRIPTION:
Chin plays an important role in the lower facial harmony and balance. With the advances in computer-aided surgical simulation (CASS) technology, surgeons are now able to simulate surgical procedures in the computer to achieve the best possible surgical plan. However, CAD/CAM surgical templates do not maximize the potential of CASS technique. Patient specific implants (PSI) has rapidly developed in cranio-maxillofacial surgery in the past few years. However, few studies have introduced PSI technique in osseous genioplasty. The purpose of this study is to assess the accuracy and clinical validation of patient specific implants (PSI) technique in genioplasty for positioning and fixation of the chin segment.

Anticipated 30 patients with chin deformities are enrolled. Virtual planning is performed with the computer-aided surgical simulation method. The 3D printing titanium cutting guide and patient specific plate is involved in this PSI method. The cutting guide is designed to guide the osteotomy and screw holes drilling for the following patient specific plate. And the patient specific plate is used to simultaneously complete the reposition and fixation of the chin. The outcome is evaluated by comparing the plan with actual outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were scheduled to undergo genioplasty;
2. patients who were scheduled to undergo CT scan as a part of their diagnosis and treatment;
3. patients who agreed to participate in this study

Exclusion Criteria:

1. craniofacial syndrome;
2. segmental osseous genioplasty;
3. previous osseous genioplasty;
4. previous mandibular trauma;
5. systemic disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Positional differences of the chin between the plan and postoperative results | 2 weeks after the operation
  The coordinates of the centroid of three land points on the chin segment was used to calculate the position differences between the plan and postoperative results in X, Y and Z axis.
Orientation differences of the chin between the plan and postoperative results | 2 weeks after the operation
  The coordinates of three independent points were used to define the orientation of the chin in 3D space. The orientation differences were calculated in pitch (the rotation around the X axis), roll (the rotation around the Y axis), and yaw (the rotation around the Z axis).

SECONDARY OUTCOMES:
time consuming | 3 days after the operation
  time spending for the virtual planning and the design of the PSI
economic consuming | 3 days after the operation
  economic cost of the fabrication of the patient specific implant

CONTACTS AND LOCATIONS:
Locations (1):
- Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided